CLINICAL TRIAL: NCT05622370
Title: An Open Label, Balanced, Randomized, 3×3 Latin Square Design Comparing of Brivaracetam Sustained-release Tablets and Brivaracetam Tablets in the Oral Comparative Pharmacokinetic(PK) Study in Chinese Healthy Adult Subjects Under Fasting Conditions.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: GX pharma technology (beijing) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GXPH-BLXTHSP-YPK
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-11

CONDITIONS: Partial Seizure
Keywords: Epilepsy; 16 years old and above; brivaracetam
MeSH Terms: conditions — Seizures; Epilepsy | interventions — brivaracetam; Tablets

STUDY DESIGN:
Intervention Model Description: Test preparation A(T1): Brivaracetam sustained-release tablets (100mg/ tablet, developed by Taizhou Overseas Pharmaceuticals Co.,Ltd.) Test preparation B(T2): Brivaracetam sustained-release tablets (50mg/ tablet, developed by Taizhou Overseas Pharmaceuticals Co.,Ltd.) Reference preparation (R): Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brivaracetam sustained-release tablets 100mg (Experimental): Brivaracetam sustained-release tablets Specification: 100mg/ tablet Batch number: 22081201 Content: 102.5% Date of production: August 12, 2022 Expiry date: August 11th, 2024. Storage conditions: sealed and stored at 10-30℃ Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Taizhou Overseas Pharmaceuticals Co.,Ltd.
  According to the random table, take test preparation A(T1) once (1 tablet/time) or test preparation B(T2) once (2 tablets/time) or reference preparation (R) twice (1 tablet/time, with an interval of 12 hours, before taking the medicine for the first time) on an empty stomach.
  Interventions: Drug: Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB); Drug: Brivaracetam sustained-release tablets 50mg
- Brivaracetam sustained-release tablets 50mg (Experimental): Brivaracetam sustained-release tablets Specification: 50mg/ piece Batch number: 22082501 Content: 100.0% Date of production: September 02, 2022 Expiry date: August 24th, 2024. Storage conditions: sealed and stored at 10-30℃ Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Taizhou Overseas Pharmaceuticals Co.,Ltd.
  According to the random table, take test preparation A(T1) once (1 tablet/time) or test preparation B(T2) once (2 tablets/time) or reference preparation (R) twice (1 tablet/time, with an interval of 12 hours, before taking the medicine for the first time) on an empty stomach.
  Interventions: Drug: Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB); Drug: Brivaracetam sustained-release tablets 100mg
- Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB) (Active Comparator): Brivaracetam tablets (trade name: Briviact) Specification: 50mg/ piece Batch number: 34244 Content: 100.0% Date of purchase: September 2022
  According to the random table, take test preparation A(T1) once (1 tablet/time) or test preparation B(T2) once (2 tablets/time) or reference preparation (R) twice (1 tablet/time, with an interval of 12 hours, before taking the medicine for the first time) on an empty stomach.
  Expiry date: April 2025 Storage conditions: sealed, stored at 20-25℃, allowing short-term temperature deviation of 15-30℃ Manufacturer: Union Chimique Belge Pharm, UCB Provider: Taizhou Overseas Pharmaceuticals Co.,Ltd.
  Interventions: Drug: Brivaracetam sustained-release tablets 100mg; Drug: Brivaracetam sustained-release tablets 50mg

INTERVENTIONS:
Drug: Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB) — Brivaracetam tablets (trade name: Briviact) Specification: 50mg/ piece Batch number: 34244 Content: 100.0% Date of purchase: September 2022
  According to the random table, take test preparation A(T1) once (1 tablet/time) or test preparation B(T2) once (2 tablets/time) or reference preparation (R) twice (1 tablet/time, with an interval of 12 hours, before taking the medicine for the first time) on an empty stomach.
  Expiry date: April 2025 Storage conditions: sealed, stored at 20-25℃, allowing short-term temperature deviation of 15-30℃ Manufacturer: Union Chimique Belge Pharm, UCB Provider: Taizhou Overseas Pharmaceuticals Co.,Ltd.
  Arms: Brivaracetam sustained-release tablets 100mg; Brivaracetam sustained-release tablets 50mg
Drug: Brivaracetam sustained-release tablets 100mg — Brivaracetam sustained-release tablets Specification: 100mg/ tablet Batch number: 22081201 Content: 102.5% Date of production: August 12, 2022 Expiry date: August 11th, 2024. Storage conditions: sealed and stored at 10-30℃ Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Taizhou Overseas Pharmaceuticals Co.,Ltd.
  According to the random table, take test preparation A(T1) once (1 tablet/time) or test preparation B(T2) once (2 tablets/time) or reference preparation (R) twice (1 tablet/time, with an interval of 12 hours, before taking the medicine for the first time) on an empty stomach.
  Arms: Brivaracetam sustained-release tablets 50mg; Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB)
Drug: Brivaracetam sustained-release tablets 50mg — Brivaracetam sustained-release tablets Specification: 50mg/ piece Batch number: 22082501 Content: 100.0% Date of production: September 02, 2022 Expiry date: August 24th, 2024. Storage conditions: sealed and stored at 10-30℃ Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Taizhou Overseas Pharmaceuticals Co.,Ltd.
  According to the random table, take test preparation A(T1) once (1 tablet/time) or test preparation B(T2) once (2 tablets/time) or reference preparation (R) twice (1 tablet/time, with an interval of 12 hours, before taking the medicine for the first time) on an empty stomach.
  Arms: Brivaracetam sustained-release tablets 100mg; Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB)

SUMMARY:
An open label, balanced, randomized, 3×3 latin square design comparing of Brivaracetam sustained-release tablets and Brivaracetam tablets in the oral comparative pharmacokinetic(PK) study in Chinese healthy adult subjects under fasting conditions.

Test preparation A(T1): Brivaracetam sustained-release tablets (100mg/ tablet, developed by Taizhou Overseas Pharmaceuticals Co.,Ltd.) Test preparation B(T2): Brivaracetam sustained-release tablets (50mg/ tablet, developed by Taizhou Overseas Pharmaceuticals Co.,Ltd.) Reference preparation (R): Brivaracetam tablets (50mg/ tablet, BRIVIACT®, UCB) Objective: The sustained-release tablets of Brivaracetam (specification: 100mg) developed by Taizhou Overseas Pharmaceuticals Co.,Ltd. were used as the test preparation A(T1), the sustained-release tablets of Brivaracetam (specification: 50mg) were used as the test preparation B(T2), and the Brivaracetam tablets (trade name: BRIVIACT®, specification: 50mg) produced by UCB were used as the reference preparation (R). To compare the blood concentration and main pharmacokinetic parameters between test preparation A(T1) and test preparation B(T2), between test preparation A(T1) and reference preparation, and between test preparation B(T2) and reference preparation, and evaluate the relative bioavailability and sustained release characteristics of test preparation.

Objective: To evaluate the safety of China healthy volunteers after oral administration of sustained-release tablets of test preparation A(T1) and B(T2) and reference preparation (R) Brivaracetam tablets on an empty stomach.

DETAILED DESCRIPTION:
Single-center, randomized, open, 3×3 Latin square design, and administration on an empty stomach. All subjects must sign an informed consent form before taking part in the trial. 12 healthy subjects (half male and half female) who passed the screening were randomly divided into three groups: T1-T2-R group, T2-R-T1 group and R-T1-T2 group, with 4 people in each group. The selected subjects entered the first ward of the clinical research center one day before taking medicine in each cycle, and fasted for more than 10 hours before taking medicine in each cycle.

On the morning of taking medicine in each cycle, after the collection of blank blood samples, the corresponding study drugs were taken according to the random table, and 240mL of warm water was taken. Eat standard lunch after 4h of the first administration, eat standard dinner after 10h, and drink water before and within 1h after the first administration (except 240mL of water used for administration). During the experiment, a unified diet is required. The test method is the same for each cycle, and the cleaning period for each cycle is 7 days.

PK blood collection and blood sample treatment:

For test preparation A(T1) and test preparation B(T2):

Before administration (0h) and 5min、10min、20min、40min、1h、1.25h、1.5h、1.75h、2h、2.5h、3h、3.5h、4h、4.5h、5h、5.5h、6h、7h、8h、10h、12h、16h、24h、36h、48h,Blood samples were collected at 26 time points.

For the reference preparation (R):

Before (0h) and after 5min、10min、20min、40min、1h、1.25h、1.5h、1.75h、2h、2.25h、2.5h、3h、4h、6h、8h、10h、12h、12.25h、12.5h、12.75h、13h、13.25h、13.5h、13.75h、14h、14.5h、15h、16h、18h、24h、36h、48h，Blood samples were collected at 33 time points.

The sitting vital signs (including body temperature, pulse and blood pressure) of the subjects were measured within 1 hour before the first administration and 2.0h±0.5h, 4.0h±0.5h, 24±1.0h and 48±1.0h after administration. In the third cycle, the subjects were examined for safety before leaving the hospital, including physical examination, vital signs examination, electrocardiogram and laboratory related examination. During the study, pay attention to observe and ask the subjects' subjective feelings and possible adverse events during the experiment. All the subjects were followed up by telephone or WeChat 7~10 days after the end of the third cycle, and asked if there were any follow-up adverse events. In case of AE, AE should be recorded and followed up.

If AE occurs during the trial, it needs to be followed up until the AE returns to normal or stable state or abnormal, which has no clinical significance or is lost.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand the purpose, nature, methods and possible adverse reactions of the experiment, volunteer as subjects, and sign an informed consent form before any research procedure starts;
2. Male and female subjects aged from 18 to 60 years (including 18 and 60 years);
3. Male weight ≥50.0 kg, female weight ≥45.0 kg, body mass index (BMI) in the range of 19.0~26.0 kg/m2 (including the critical value);
4. The subject has no history of chronic diseases or serious diseases such as cardiovascular, liver, kidney, blood and lymph, endocrine, immune, mental, nervous, gastrointestinal system, etc., and is in good general health;
5. During screening, vital signs examination, physical examination, clinical laboratory examination (blood routine examination, urine routine examination, blood biochemistry examination, hepatitis B, hepatitis C, AIDS and syphilis examination, coagulation function), pregnancy examination (only for women), chest X-ray examination, 12-lead electrocardiogram and nicotine examination, the results show that there is no abnormality or no clinical significance;
6. Subjects (including male subjects) have no pregnancy plans and voluntarily take effective contraceptive measures from two weeks before the screening date to six months after the last administration, and have no plans for sperm donation or egg donation; Female subjects/male subjects and their female partners of childbearing age did not have unprotected sex within one month before the screening, and female subjects agreed not to use contraceptives from the screening to the end of the trial;
7. Subjects can communicate well with researchers, and understand and abide by the requirements of this research.

Exclusion Criteria:

1. those who have a history of allergy to research drugs or their adjuvants, or are allergic to drugs, food, pollen or have a specific history of allergy (asthma, allergic rhinitis, eczema), etc.;
2. Have a history of dysphagia or any gastrointestinal diseases that affect drug absorption;
3. Anyone who has a history of surgery or trauma that may affect the safety of the trial or the in vivo process of the drug, or who plans to have surgery during the study period;
4. Any prescription drugs, over-the-counter drugs, Chinese herbal medicines and health products were taken orally within 28 days before the screening, especially any drugs that change the activity of liver enzymes (such as: inducers-barbiturates, carbamazepine, phenytoin, glucocorticoid, omeprazole; Inhibitors--SSRI antidepressants, cimetidine, diltiazem macrocyclic lipids, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines, etc.);
5. Screening those who have a history of drug abuse within 6 months before;
6. Screening those who have used drugs within the first 3 months;
7. Screening those who have been vaccinated within 2 months before screening;
8. Those who smoke more than 5 cigarettes per day within 3 months before screening, or can't stop using any tobacco products during the trial period;
9. Drinking more than 14 units per week (1 unit = 17.7 mL of ethanol, that is, 1 unit = 357 mL of 5% alcohol beer or 43 mL of 40% alcohol liquor or 147 mL of 12% alcohol wine) within 3 months before screening, or those who can't abstain from drinking during the experiment;
10. Those who drink excessive tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250 ml) every day within 3 months before screening;
11. those who have participated in other drug clinical trials within 3 months before administration or who have not participated in clinical trials by themselves;
12. Blood donation within 3 months before screening includes blood component or massive blood loss (≥450mL), and those who receive blood transfusion or use blood products are planned to donate blood during the test period;
13. The subject (female) is in lactation;
14. Those who can't tolerate venipuncture and have a history of fainting from needles and blood;
15. Those who have special requirements for diet and cannot accept a unified diet;
16. Screening those who have had significantly abnormal diet (such as dieting and low sodium) within 1 month before screening;
17. Subjects judged by other researchers to be unsuitable for participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma concentration of the period (AUC0-last) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | 1 month
  Individual Brivaracetam plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual brivaracetam plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual brivaracetam plasma concentration-time profile for each treatment period will be established.
Mean residence time (MRT) | 1 month
  Individual brivaracetam plasma concentration-time profile for each treatment period will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Municipal People's Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No